CLINICAL TRIAL: NCT01594762
Title: A Randomized, Double-Blind, Multicenter, Superiority, Placebo-Controlled Phase 3 Study of Pexiganan Cream 0.8% Applied Twice Daily for 14 Days in the Treatment of Adults With Mild Infections of Diabetic Foot Ulcers
Brief Title: Pexiganan Versus Placebo Control for the Treatment of Mild Infections of Diabetic Foot Ulcers
Acronym: OneStep-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dipexium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DPX-306
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Foot Infection
Keywords: Diabetic Foot Ulcer Infection
MeSH Terms: interventions — pexiganan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topical placebo control (Placebo Comparator): Drug: Topical placebo cream
  Interventions: Drug: Topical placebo cream; Other: Standard wound care
- Topical pexiganan cream 0.8% (Experimental): Drug: Topical pexiganan cream 0.8%
  Interventions: Drug: Topical pexiganan cream 0.8%; Other: Standard wound care

INTERVENTIONS:
Drug: Topical pexiganan cream 0.8% — 14 days of treatment
  Other Names: MSI-78
  Arms: Topical pexiganan cream 0.8%
Drug: Topical placebo cream — 14 days of treatment
  Arms: Topical placebo control
Other: Standard wound care — 14 days of treatment

SUMMARY:
The purpose of this study is to establish the clinical superiority and the safety of topical pexiganan cream 0.8% plus standard local wound care as compared to placebo cream plus standard local wound care, in the treatment of mildly infected diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus.
2. Male or female at least 18 years old.
3. Subject must agree to adhere to all protocol procedures and return for all scheduled visits, and must be willing and able to provide written informed consent.
4. Subject is to be treated on an outpatient basis.
5. Full thickness ulcer or a partial thickness ulcer on the foot distal to the malleoli with a surface area ≥ 1 cm2 after the wound has undergone appropriate debridement.
6. Localized mild infection of the ulcer.
7. The diagnosis of mild infection must be confirmed immediately following debridement at Baseline.
8. Subject must have plain radiographs taken within 2 days prior to entry showing no evidence of bony abnormalities consistent with osteomyelitis, or gas compatible with tissue crepitus, in the affected foot.

Exclusion Criteria:

1. IDSA-defined moderate infection, including cellulitis extending > 2 cm; lymphangitis; spread beneath the fascia; deep tissue abscess; gangrene; muscle, joint, or bone involvement.
2. IDSA-defined severe infection, including systemic toxicity or metabolic instability.
3. Infected diabetic foot ulcer that is associated with local wound complications such as prosthetic materials or protruding surgical hardware.
4. > 1 infected foot ulcer.
5. Subject is currently receiving topical antimicrobial treatment for a localized infection of the study ulcer and whose infection is improving in response to treatment.
6. Subject has received a systemic antibiotic within 48 hours prior to Screening.
7. Concurrent or expected to require systemic antimicrobials during the study period for any infection, including diabetic foot ulcer.
8. Bone or joint involvement is suspected based on clinical examination or plain X-ray.
9. Clinically significant peripheral arterial disease requiring vascular intervention.
10. Subject is expected to be unable to care for the ulcer or return for all scheduled visits because of hospitalization, vacation, disability, etc. during the study period, or is unable to safely monitor the infection status at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Silverman, MD, Study Director — Biostrategics Consulting Ltd
Locations (39):
- United States (39):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Castro Valley, California
  - Davis, California
  - Los Angeles, California
  - Napa, California
  - San Francisco, California
  - Santa Rosa, California
  - Sylmar, California
  - Vacaville, California
  - Norwalk, Connecticut
  - Coral Gables, Florida
  - Doral, Florida
  - Hialeah, Florida
  - Homestead, Florida
  - Jacksonville, Florida
  - Largo, Florida
  - Miami, Florida
  - Miami Lakes, Florida
  - Miami Shores, Florida
  - Pinellas Park, Florida
  - Evans, Georgia
  - North Chicago, Illinois
  - Hutchinson, Kansas
  - New Orleans, Louisiana
  - Mineola, New York
  - Charlotte, North Carolina
  - Wilmington, North Carolina
  - Duncansville, Pennsylvania
  - York, Pennsylvania
  - Columbia, South Carolina
  - El Paso, Texas
  - Fort Worth, Texas
  - Lewisville, Texas
  - Salt Lake City, Utah
  - St. George, Utah
  - Roanoke, Virginia
  - Richland, Washington

REFERENCES:
- [Derived] You Y, Liu H, Zhu Y, Zheng H. Rational design of stapled antimicrobial peptides. Amino Acids. 2023 Apr;55(4):421-442. doi: 10.1007/s00726-023-03245-w. Epub 2023 Feb 12. PMID 36781451

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Pexiganan Cream 0.8%: Drug: Topical pexiganan cream 0.8%
  Topical pexiganan cream 0.8%: 14 days of treatment + 14 days of follow-up (28-day trial period)
  Standard wound care: 28-day trial period
- Topical Placebo Control: Drug: Topical placebo cream
  Topical placebo cream: 14 days of treatment + 14 days of follow-up (28-day trial period)
  Standard wound care: 28-day trial period
Period: Overall Study
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Started | 97 | 103
Completed | 86 | 93
Not Completed | 11 | 10
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Topical Pexiganan Cream 0.8%: Drug: Topical pexiganan cream 0.8%
  Topical pexiganan cream 0.8%: 14 days of treatment
  Standard wound care: 28-day trial period
- Topical Placebo Control: Drug: Topical placebo cream
  Topical placebo cream: 14 days of treatment
  Standard wound care: 28-day trial period
- Total: Total of all reporting groups
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control | Total
Number analyzed (Participants) | 97 | 103 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.37 (12.71) | 57.14 (10.61) | 57.25 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 70 | 81 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 35 | 66
  Not Hispanic or Latino | 66 | 68 | 134
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 27 | 46
  White | 78 | 75 | 153
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 97 | 103 | 200
Wound surface area [Count of Participants; unit: Participants]
  <1 sq cm | 4 | 5 | 9
  1 - <2 sq cm | 50 | 54 | 104
  >=2 sq cm | 43 | 43 | 86
  Missing | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response
Description: The numbers of participants with Clinical Response, defined as resolution of infection, are reported.
Time Frame: 28 days
Population: Intent-To-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Number analyzed (Participants) | 97 | 103
Participants | 56 | 54

2. Secondary Outcome: Number of Participants With Microbiological Response
Description: The numbers of participants with Microbiological Response, defined are eradication of all baseline pathogens, are reported.
Time Frame: 28 days
Population: Intent-To-Treat Microbiological (positive for baseline pathogens)
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Number analyzed (Participants) | 63 | 75
Participants | 18 | 27

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: The number of participants with TEAEs, including Serious TEAEs, are reported
Time Frame: 28 days
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
Number analyzed (Participants) | 97 | 103
Participants
  Incidence of any TEAE | 25 | 21
  Incidence of Serious TEAE | 8 | 2

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Topical Pexiganan Cream 0.8% | Topical Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/103
Serious Adverse Events (participants affected / at risk) | 8/97 | 2/103
Other Adverse Events (participants affected / at risk) | 6/97 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Pexiganan Cream 0.8% (N=97) | Topical Placebo Control (N=103)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (1)
Diabetic ketoacidiosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Foot surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Pexiganan Cream 0.8% (N=97) | Topical Placebo Control (N=103)
Osteomyelitis (Infections and infestations) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no multi-site publication within 18 months of study completion, Site shall have right to publish subject to: 1) Prior to submitting/presenting, Site shall provide Sponsor a copy; Sponsor shall have 60 days to review/comment. 2) Site shall remove any Confidential Information prior to submitting/presenting the materials. 3) Site shall further delay publication/presentation for up to 120 days to allow Sponsor to protect its interests in any Sponsor Inventions described in any such materials.